CLINICAL TRIAL: NCT00388362
Title: A Phase II Trial of Sirolimus as Treatment of Steroid-Refractory or Steroid-Dependent Chronic Graft-Versus-Host Disease
Brief Title: Sirolimus as Treatment of Steroid-Refractory or Steroid-Dependent Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura Johnston, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-3587; 96589 (Other: Stanford University Alternate IRB Approval Number); BMT175 (Other: OnCore Number)
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Graft vs Host Disease
Keywords: GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus Therapy (Experimental): Administration of Sirolimus and Prednisone
  Interventions: Drug: Sirolimus; Drug: Prednisone

INTERVENTIONS:
Drug: Sirolimus — Patients will receive sirolimus at 2 mg/day orally with monitoring of trough drug levels weekly for 2 weeks to achieve trough drug levels 7-12 ng/ml. Along with prednisone therapy.
  Other Names: Rapamune
Drug: Prednisone — Prednisone therapy will remain at the dose the patient received at the time sirolimus was begun. Withdrawal of prednisone will began after first evidence of improvement of chronic GVHD.
  Other Names: Deltasone

SUMMARY:
To study the effectiveness of an immunosuppressive drug sirolimus, in the treatment of chronic graft versus host disease in combination with prednisone.

DETAILED DESCRIPTION:
The purpose of this trial is to study the effectiveness of an immunosuppressive drug, sirolimus, in the treatment of chronic graft versus host disease in combination with prednisone. Graft versus host disease (GVHD) is a common complication in patients who have received blood or marrow transplantation from a related or unrelated donor. Chronic GVHD occurs approximately 100 days after transplantation and is the result of the donor immune system recognizing the patient's tissues as foreign and creating harmful effects on the patient's organs. We hope the use of sirolimus will decrease the significant disabling effects and deaths caused by chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 13 years
* Weight ≥ 40 kg.
* Biopsy or clinical presentation diagnostic of chronic GVHD >100 days following allogeneic bone marrow/peripheral blood/umbilical cord blood transplantation that has failed prior corticosteroid therapy or corticosteroid taper. In the event that histological confirmation poses undue risk, clinical evaluation is sufficient.
* Women of child-bearing potential must have a negative pregnancy test before sirolimus administration and agree to use a medically acceptable contraceptive throughout the treatment period until 3 months after discontinuation of sirolimus.
* Any woman becoming pregnant during the treatment period must discontinue the use of sirolimus.
* Absolute neutrophil count (ANC) > 1000/mm³, unless receiving G-CSF to maintain neutrophil count > 500/mm³.
* At the time of initiating sirolimus the cyclosporine trough level is recommended to be < 100 mg/dl and FK506 level is recommended to be < 5 mg/dl. FK506 or cyclosporine is to be discontinued soon after initiation of sirolimus.
* Karnofsky performance score ≥ 50 during pre-study screening.
* Written, signed, and dated informed consent

Exclusion Criteria:

* Uncontrolled systemic infection
* Unstable disease states (i.e., hepatic failure, ventilatory-dependent respiratory failure, etc.)
* Serum creatinine ≥ 3.0 mg/dL
* Platelet count ≤ 50,000/mm³
* History of Post-transplant microangiopathic hemolytic anemia
* Uncontrolled hyperlipidemia
* Use of any investigational drug within 4 weeks of entry into the study
* Use of methotrexate or antibody therapies within 24 hours of sirolimus administration
* Inability to tolerate oral therapy for any reason
* Evidence of infiltrate, cavitation, or consolidation on chest x-ray during pre-study screening
* Known hypersensitivity to macrolide antibiotics

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-11; Primary Completion 2010-11 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnston, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Enrolled
Arm/Group | Sirolimus Therapy
Started | 36
Completed | 23
Not Completed | 13
Not completed — Ineligible | 1
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Loss insurance | 1
Not completed — Withdrawal by Subject | 1
Period: Remained on Study Median of 514 Days
Arm/Group | Sirolimus Therapy
Started | 23
Completed | 21
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Administration of Sirolimus and Prednisone
Groups:
- Sirolimus: Administration of Sirolimus and Prednisone
Arm/Group | Sirolimus
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Activity
Description: Determined by discontinuation of immunosuppression with resolution of all reversible CGVHD manifestations. Evaluated at 2 years after enrollment
Time Frame: 3 month intervals after the initiation of sirolimus until 2 years after the initiation of sirolimus
Population: 23 patients that remained on the study for a median of 514 days (96-814 days). Numbers based on resolution/ improvement in clinical manifestations of cGVHD with a median of 90% reduction in prednisone dose and no additional immunosuppressive therapy over a two year treatment period.
Measure: Number; unit: participants
Arm/Group | Sirolimus Therapy
Number analyzed (Participants) | 23
participants
  Complete Remission | 4
  Partial Remission | 4

2. Secondary Outcome: Overall Survival
Description: Administration of Sirolimus and Prednisone
Time Frame: 3 month intervals after the initiation of sirolimus until 2 years after the initiation of sirolimus
Population: 23 patients that remained on the study for a median of 514 days (96-814 days), 2 died (1- second cancer and 1- progressive cardiac failure)
Measure: Number; unit: participants
Arm/Group | Sirolimus Therapy
Number analyzed (Participants) | 23
participants | 21

ADVERSE EVENTS:
Time Frame: 2 years after enrollment
Arm/Group | Sirolimus Therapy
Serious Adverse Events (participants affected / at risk) | 14/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Therapy (N=35)
Death (General disorders) | 1 (1)
CMV resulting in death (Infections and infestations) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sirolimus associated interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sirolimus associated thrombotic microangiopathy and hypertriglyceridemia resulting in pancreatitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematological Disease Relapse (Blood and lymphatic system disorders) | 2 (2)
Emergent Surgery (General disorders) | 1 (1)
Metapneumovirus pneumonia, recurrent PE resulting in death (Infections and infestations) | 1 (1)
Recurrent Viral Pneumonia (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Therapy (N=35)
Infection (Infections and infestations) | 15 (15) — Any infection
Edema (Musculoskeletal and connective tissue disorders) | 8 (8) — Limb
Cholesterol (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
hypertriglyceridema (Blood and lymphatic system disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No